CLINICAL TRIAL: NCT00005049
Title: Pilot Study of Intraperitoneal (IP) Therapy With Cisplatin or Carboplatin and Floxuridine (FUdR) as Consolidation for Ovarian and Gastrointestinal Malignancies
Brief Title: Combination Chemotherapy in Treating Patients With Stage III Ovarian Epithelial Cancer or Gastrointestinal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067641; P30CA016087 (NIH); NYU-9645; NCI-G00-1717
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Colorectal Cancer; Gastric Cancer; Gastrointestinal Carcinoid Tumor; Gastrointestinal Stromal Tumor; Ovarian Cancer; Peritoneal Cavity Cancer; Small Intestine Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage II gastric cancer; stage III gastric cancer; recurrent gastric cancer; stage II rectal cancer; stage III rectal cancer; recurrent colon cancer; stage III ovarian epithelial cancer; recurrent ovarian epithelial cancer; regional gastrointestinal carcinoid tumor; small intestine adenocarcinoma; small intestine lymphoma; small intestine leiomyosarcoma; recurrent small intestine cancer; peritoneal cavity cancer; gastrointestinal stromal tumor
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Gastrointestinal Stromal Tumors; Ovarian Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cisplatin; Floxuridine

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: floxuridine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving them by intraperitoneal infusion may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of intraperitoneal combination chemotherapy in treating patients who have stage III ovarian epithelial cancer or gastrointestinal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess tolerance and complications from consolidation therapy with intraperitoneal floxuridine and cisplatin and/or carboplatin in patients with stage III ovarian epithelial cancer or gastrointestinal cancer with peritoneal involvement.
* Determine the sites of failure and estimate the time to failure following treatment with this regimen in these patients.

OUTLINE: Patients are stratified according to type of residual disease at second look laparotomy or laparoscopy (micro only vs no greater than 0.5 cm vs greater than 0.5 cm and no greater than 1 cm), and by CA-125 level (elevated vs normal on day -7).

Patients receive intraperitoneal floxuridine on days 1-3 followed by intraperitoneal cisplatin and/or carboplatin on day 3. Treatment continues every 3 weeks for 4-6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 and 6 weeks, then at 6, 12, 18, and 24 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage III ovarian epithelial cancer or gastrointestinal cancer with peritoneal involvement
* Patients with ovarian cancer must have completed first induction treatment with a platinum based regimen (carboplatin and/or cisplatin) and be in clinical complete response at time of assessment for study
* No ovarian cancer of low malignant potential

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Greater than 2 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT less than 3 times upper limit of normal

Renal:

* Creatinine clearance at least 40 mL/min

Other:

* No underlying medical or psychiatric condition that precludes informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Laparoscopy or laparotomy required within 8 weeks of study to assess residual disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1997-05; Primary Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States